CLINICAL TRIAL: NCT01039350
Title: Prospective, Multicenter, Open Label and Single-arm Study of Darbepoetin Alfa for Anemia in Myelodisplastic Syndrome Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was stopped due to a lack of recruitment after 48 patients included
Sponsor: Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon (Other)
Responsible Party: Ana M Villegas, FEHH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEE200401; 2005-002414-38 (EudraCT Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa will be initiated at a weekly (QW) subcutaneous dose of 300 mcg over 8 weeks.

SUMMARY:
This is an open-label, single-arm, multicentre, prospective study of darbepoetin alfa to treat anaemia in patients with low and intermediate-1 IPSS risk MDS. The study will consist of a 14-day screening period followed by a maximum 24-week treatment period and a final visit.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicentre, prospective study of darbepoetin alfa to treat anaemia in patients with low and intermediate-1 IPSS risk MDS. The study will consist of a 14-day screening period followed by a maximum 24-week treatment period and a final visit. Darbepoetin alfa will be initiated at a dose of 300 mcg QW SC over a period of 8 weeks. After 8 weeks, erythroid response will be evaluated, and treatment algorithm adapted to it.

The study treatment period will last for a maximum of 24 weeks. The treatment will end at the start of week 24. If the scheduled 24-week treatment period is not completed, it will end during the week of the last administration of the study drug.

The follow-up period will last for a minimum of 4 weeks and a maximum of 8 weeks after the last dose of darbepoetin alfa.

Subjects will be stratified at enrolment according to IPSS (low risk versus intermediate-1 risk).

ELIGIBILITY:
Inclusion Criteria:

* Age ³ 18 years
* Low or intermediate-1 risk MDS according to IPSS, and FAB classification of RA, RARS, or RAEB with blasts £ 10%
* Predictive variables of good response (serum erythropoietin levels < 500 IU/l and transfusion requirements < 2 packed RBC/month over the preceding 2 months)
* Anaemia (Hb £ 10 g/dL), confirmed in the 14 days before day 1 of the study
* Life expectancy of at least 6 months
* ECOG Performance status score of 0, 1, or 2
* Subject must sign and date the Informed Consent (approved by a Clinical Research Ethics Committee - CREC), before any study-specific procedure is performed

Exclusion Criteria:

* Known history of convulsive disorders
* Poorly controlled hypertension (diastolic blood pressure > 100 mmHg) at screening
* Inadequate liver function (total bilirubin > two times the upper limit of the normal range (ULN), and liver enzymes (ALT, AST) > two times ULN)
* Inadequate renal function (serum creatinine concentration > 2 mg/dL)
* Ferritin < 100 ng/ml or transferrin saturation index (TSI) < 16%; Vitamin B12 deficiency (< 200 pg/ml) or folate deficiency (< 2 ng/ml)
* Clinically-relevant haemorrhages
* Haemolytic anaemia
* Cardiac condition: uncontrolled angina, congestive heart failure, or uncontrolled cardiac arrhythmia
* Clinically significant systemic infection or chronic inflammatory disease present at time of screening
* Any concomitant therapy used to treat MDS (including other growth factors than those described as part of this protocol, chemotherapy, antibody-based cancer treatment, hormonal therapy, interferon, and interleukins)
* Treatment with rHuEPO or darbepoetin alfa over the 4 weeks prior to Day 1 of the study
* More than 2 RBC transfusions over the 28 days prior to Day 1 of the study
* Pregnant or breast feeding women
* Subjects of childbearing-potential who do not take adequate contraceptive measures, in the opinion of the investigator
* Known hypersensitivity to any mammal-derived recombinant product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving an erythroid response during the 24-week treatment period. | weeks 8; 12; 16 and 24

SECONDARY OUTCOMES:
Time to erythroid response and time it is maintained. | week 24
Proportion of non-responders to darbepoetin alfa who obtain an erythroid response after the addition of Filgrastim | weeks 8, 12, 16 and 24
Proportion of patients receiving RBC transfusions (more than 1 unit) from week 5 to 24, inclusive | weeks 8; 12; 16 and 24
Score changes in the FACT-Fatigue quality-of-life scale between the baseline visit, and weeks 8, 16, 24, and the end of the study. | weeks 8; 16 and 24
Number of morphological and cytogenetic disorders at baseline and end of treatment | week 24
Incidence of adverse events and serious adverse events | weeks 8; 12; 16 and 24
Proportion of patients with haemoglobin values over 12 g/dL at any time during the study | weeks 8; 12; 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Villegas, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon
Locations (16):
- Spain (16):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Vall D´Hebron, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona, Barcelona
  - Hospital de Cruces, Barakaldo, Bilbao
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital Virgen del Puerto, Plasencia, Caceres
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Universitario Juan Canalejo, A Coruña, La Coruña
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario La Fé, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia

REFERENCES:
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] Nosslinger T, Reisner R, Koller E, Gruner H, Tuchler H, Nowotny H, Pittermann E, Pfeilstocker M. Myelodysplastic syndromes, from French-American-British to World Health Organization: comparison of classifications on 431 unselected patients from a single institution. Blood. 2001 Nov 15;98(10):2935-41. doi: 10.1182/blood.v98.10.2935. PMID 11698274
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Littlewood TJ. Erythropoietin for the treatment of anemia associated with hematological malignancy. Hematol Oncol. 2001 Mar;19(1):19-30. doi: 10.1002/hon.663. PMID 11276043
- [Background] Molldrem JJ, Leifer E, Bahceci E, Saunthararajah Y, Rivera M, Dunbar C, Liu J, Nakamura R, Young NS, Barrett AJ. Antithymocyte globulin for treatment of the bone marrow failure associated with myelodysplastic syndromes. Ann Intern Med. 2002 Aug 6;137(3):156-63. doi: 10.7326/0003-4819-137-3-200208060-00007. PMID 12160363
- [Background] Raza A, Meyer P, Dutt D, Zorat F, Lisak L, Nascimben F, du Randt M, Kaspar C, Goldberg C, Loew J, Dar S, Gezer S, Venugopal P, Zeldis J. Thalidomide produces transfusion independence in long-standing refractory anemias of patients with myelodysplastic syndromes. Blood. 2001 Aug 15;98(4):958-65. doi: 10.1182/blood.v98.4.958. PMID 11493439
- [Background] Stasi R, Pagano A, Terzoli E, Amadori S. Recombinant human granulocyte-macrophage colony-stimulating factor plus erythropoietin for the treatment of cytopenias in patients with myelodysplastic syndromes. Br J Haematol. 1999 Apr;105(1):141-8. PMID 10233377
- [Background] Negrin RS, Stein R, Doherty K, Cornwell J, Vardiman J, Krantz S, Greenberg PL. Maintenance treatment of the anemia of myelodysplastic syndromes with recombinant human granulocyte colony-stimulating factor and erythropoietin: evidence for in vivo synergy. Blood. 1996 May 15;87(10):4076-81. PMID 8639764
- [Background] Koury MJ, Bondurant MC. The molecular mechanism of erythropoietin action. Eur J Biochem. 1992 Dec 15;210(3):649-63. doi: 10.1111/j.1432-1033.1992.tb17466.x. No abstract available. PMID 1483451
- [Background] Rigolin GM, Porta MD, Bigoni R, Cavazzini F, Ciccone M, Bardi A, Cuneo A, Castoldi G. rHuEpo administration in patients with low-risk myelodysplastic syndromes: evaluation of erythroid precursors' response by fluorescence in situ hybridization on May-Grunwald-Giemsa-stained bone marrow samples. Br J Haematol. 2002 Dec;119(3):652-9. doi: 10.1046/j.1365-2141.2002.03867.x. PMID 12437640
- [Background] Hellstrom-Lindberg E, Ahlgren T, Beguin Y, Carlsson M, Carneskog J, Dahl IM, Dybedal I, Grimfors G, Kanter-Lewensohn L, Linder O, Luthman M, Lofvenberg E, Nilsson-Ehle H, Samuelsson J, Tangen JM, Winqvist I, Oberg G, Osterborg A, Ost A. Treatment of anemia in myelodysplastic syndromes with granulocyte colony-stimulating factor plus erythropoietin: results from a randomized phase II study and long-term follow-up of 71 patients. Blood. 1998 Jul 1;92(1):68-75. PMID 9639501
- [Background] Remacha AF, Arrizabalaga B, Villegas A, Manteiga R, Calvo T, Julia A, Fernandez Fuertes I, Gonzalez FA, Font L, Junca J, del Arco A, Malcorra JJ, Equiza EP, de Mendiguren BP, Romero M. Erythropoietin plus granulocyte colony-stimulating factor in the treatment of myelodysplastic syndromes. Identification of a subgroup of responders. The Spanish Erythropathology Group. Haematologica. 1999 Dec;84(12):1058-64. PMID 10586205
- [Background] Thompson JA, Gilliland DG, Prchal JT, Bennett JM, Larholt K, Nelson RA, Rose EH, Dugan MH. Effect of recombinant human erythropoietin combined with granulocyte/ macrophage colony-stimulating factor in the treatment of patients with myelodysplastic syndrome. GM/EPO MDS Study Group. Blood. 2000 Feb 15;95(4):1175-9. PMID 10666187
- [Background] Hast R, Wallvik J, Folin A, Bernell P, Stenke L. Long-term follow-up of 18 patients with myelodysplastic syndromes responding to recombinant erythropoietin treatment. Leuk Res. 2001 Jan;25(1):13-18. doi: 10.1016/s0145-2126(00)00073-4. PMID 11137555
- [Background] Italian Cooperative Study Group for rHuEpo in Myelodysplastic Syndromes; Ferrini PR, Grossi A, Vannucchi AM, Barosi G, Guarnone R, Piva N, Musto P, Balleari E. A randomized double-blind placebo-controlled study with subcutaneous recombinant human erythropoietin in patients with low-risk myelodysplastic syndromes. Br J Haematol. 1998 Dec;103(4):1070-4. doi: 10.1046/j.1365-2141.1998.01085.x. PMID 9886322
- [Background] Terpos E, Mougiou A, Kouraklis A, Chatzivassili A, Michalis E, Giannakoulas N, Manioudaki E, Lazaridou A, Bakaloudi V, Protopappa M, Liapi D, Grouzi E, Parharidou A, Symeonidis A, Kokkini G, Laoutaris NP, Vaipoulos G, Anagnostopoulos NI, Christakis JI, Meletis J, Bourantas KL, Zoumbos NC, Yataganas X, Viniou NA; Greek MDS Study Group. Prolonged administration of erythropoietin increases erythroid response rate in myelodysplastic syndromes: a phase II trial in 281 patients. Br J Haematol. 2002 Jul;118(1):174-80. doi: 10.1046/j.1365-2141.2002.03583.x. PMID 12100145
- [Background] Hellstrom-Lindberg E. Efficacy of erythropoietin in the myelodysplastic syndromes: a meta-analysis of 205 patients from 17 studies. Br J Haematol. 1995 Jan;89(1):67-71. doi: 10.1111/j.1365-2141.1995.tb08909.x. PMID 7833279
- [Background] Mantovani L, Lentini G, Hentschel B, Wickramanayake PD, Loeffler M, Diehl V, Tesch H. Treatment of anaemia in myelodysplastic syndromes with prolonged administration of recombinant human granulocyte colony-stimulating factor and erythropoietin. Br J Haematol. 2000 May;109(2):367-75. doi: 10.1046/j.1365-2141.2000.02016.x. PMID 10848827
- [Background] Casadevall N, Durieux P, Dubois S, Hemery F, Lepage E, Quarre MC, Damaj G, Giraudier S, Guerci A, Laurent G, Dombret H, Chomienne C, Ribrag V, Stamatoullas A, Marie JP, Vekhoff A, Maloisel F, Navarro R, Dreyfus F, Fenaux P. Health, economic, and quality-of-life effects of erythropoietin and granulocyte colony-stimulating factor for the treatment of myelodysplastic syndromes: a randomized, controlled trial. Blood. 2004 Jul 15;104(2):321-7. doi: 10.1182/blood-2003-07-2252. Epub 2004 Mar 30. PMID 15054036
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Hellstrom-Lindberg E, Gulbrandsen N, Lindberg G, Ahlgren T, Dahl IM, Dybedal I, Grimfors G, Hesse-Sundin E, Hjorth M, Kanter-Lewensohn L, Linder O, Luthman M, Lofvenberg E, Oberg G, Porwit-MacDonald A, Radlund A, Samuelsson J, Tangen JM, Winquist I, Wisloff F; Scandinavian MDS Group. A validated decision model for treating the anaemia of myelodysplastic syndromes with erythropoietin + granulocyte colony-stimulating factor: significant effects on quality of life. Br J Haematol. 2003 Mar;120(6):1037-46. doi: 10.1046/j.1365-2141.2003.04153.x. PMID 12648074
- [Background] Egrie JC, Browne JK. Development and characterization of novel erythropoiesis stimulating protein (NESP). Br J Cancer. 2001 Apr;84 Suppl 1(Suppl 1):3-10. doi: 10.1054/bjoc.2001.1746. PMID 11308268
- [Background] Smith R. Applications of darbepoietin-alpha, a novel erythropoiesis-stimulating protein, in oncology. Curr Opin Hematol. 2002 May;9(3):228-33. doi: 10.1097/00062752-200205000-00009. PMID 11953669
- [Background] Macdougall IC, Gray SJ, Elston O, Breen C, Jenkins B, Browne J, Egrie J. Pharmacokinetics of novel erythropoiesis stimulating protein compared with epoetin alfa in dialysis patients. J Am Soc Nephrol. 1999 Nov;10(11):2392-5. doi: 10.1681/ASN.V10112392. PMID 10541299
- [Background] Kotasek D, Steger G, Faught W, Underhill C, Poulsen E, Colowick AB, Rossi G, Mackey J; Aranesp 980291 Study Group. Darbepoetin alfa administered every 3 weeks alleviates anaemia in patients with solid tumours receiving chemotherapy; results of a double-blind, placebo-controlled, randomised study. Eur J Cancer. 2003 Sep;39(14):2026-34. doi: 10.1016/s0959-8049(03)00456-8. PMID 12957457
- [Background] Hellstrom-Lindberg E, Negrin R, Stein R, Krantz S, Lindberg G, Vardiman J, Ost A, Greenberg P. Erythroid response to treatment with G-CSF plus erythropoietin for the anaemia of patients with myelodysplastic syndromes: proposal for a predictive model. Br J Haematol. 1997 Nov;99(2):344-51. doi: 10.1046/j.1365-2141.1997.4013211.x. PMID 9375752
- [Background] Glaspy JA, Jadeja JS, Justice G, Kessler J, Richards D, Schwartzberg L, Tchekmedyian NS, Armstrong S, O'Byrne J, Rossi G, Colowick AB. Darbepoetin alfa given every 1 or 2 weeks alleviates anaemia associated with cancer chemotherapy. Br J Cancer. 2002 Jul 29;87(3):268-76. doi: 10.1038/sj.bjc.6600465. PMID 12177793
- [Background] Musto P, Lanza F, Balleari E, Grossi A, Falcone A, Sanpaolo G, Bodenizza C, Scalzulli PR, La Sala A, Campioni D, Ghio R, Cascavilla N, Carella AM. Darbepoetin alpha for the treatment of anaemia in low-intermediate risk myelodysplastic syndromes. Br J Haematol. 2005 Jan;128(2):204-9. doi: 10.1111/j.1365-2141.2004.05288.x. PMID 15638854
- [Background] Mannone L, Gardin C, Quarre MC, Bernard JF, Vassilieff D, Ades L, Park S, Vaultier S, Hamza F, Beyne-rauzy MO, Cheze S, Giraudier S, Agape P, Legros L, Voillat L, Dreyfus F, Fenaux P; Groupe Francais des Myelodysplasies. High-dose darbepoetin alpha in the treatment of anaemia of lower risk myelodysplastic syndrome results of a phase II study. Br J Haematol. 2006 Jun;133(5):513-9. doi: 10.1111/j.1365-2141.2006.06070.x. PMID 16681638
- [Background] Vansteenkiste J, Pirker R, Massuti B, Barata F, Font A, Fiegl M, Siena S, Gateley J, Tomita D, Colowick AB, Musil J; Aranesp 980297 Study Group. Double-blind, placebo-controlled, randomized phase III trial of darbepoetin alfa in lung cancer patients receiving chemotherapy. J Natl Cancer Inst. 2002 Aug 21;94(16):1211-20. doi: 10.1093/jnci/94.16.1211. PMID 12189224
- [Background] Hedenus M, Adriansson M, San Miguel J, Kramer MH, Schipperus MR, Juvonen E, Taylor K, Belch A, Altes A, Martinelli G, Watson D, Matcham J, Rossi G, Littlewood TJ; Darbepoetin Alfa 20000161 Study Group. Efficacy and safety of darbepoetin alfa in anaemic patients with lymphoproliferative malignancies: a randomized, double-blind, placebo-controlled study. Br J Haematol. 2003 Aug;122(3):394-403. doi: 10.1046/j.1365-2141.2003.04448.x. PMID 12877666
- [Background] Smith RE Jr, Tchekmedyian NS, Chan D, Meza LA, Northfelt DW, Patel R, Austin M, Colowick AB, Rossi G, Glaspy J. A dose- and schedule-finding study of darbepoetin alpha for the treatment of chronic anaemia of cancer. Br J Cancer. 2003 Jun 16;88(12):1851-8. doi: 10.1038/sj.bjc.6600994. PMID 12799626
- [Background] Hellstrom-Lindberg E. Growth factor treatment for the anemia of MDS: mechanisms and efficacy. Educational Programme at the 8th Congress of the European Haematology Association (EHA), June 2003
- [Background] Verhoef GEG, Boogaerts MA. RHuEPO in the treatment of the myelodysplastic syndromes. In: Smyth JF, Boogaerts MA, Ehmer BR-M (eds): rHuEPO in cancer supportive treatment. Marcel Dekker, New York 1996;pp.13-34.
- [Background] Heatherington AC, Schuller J, Kotasek D, et al. The pharmacokinetics of darbepoetin alfa and changes in endogenous erythropoietin in patients with nonmyeloid malignancies receiving or not receiving chemotherapy. European Breast Cancer Conference (EBCC) 2002. Abstract.
- [Background] Glaspy J, Appelbaum S, Henry D et al. Effects of darbepoetin alfa (Aranesp®) timing with chemotherapy administration: a randomized study. SIOG 2003. Poster.
- [Background] WHO Classification Tumours of Haematopoietic and Lymphoid Tissues. IARC Press, Lyon 2001
- [Derived] Villegas A, Arrizabalaga B, Fernandez-Lago C, Castro M, Mayans JR, Gonzalez-Porras JR, Duarte RF, Remacha AF, Luno E, Gasquet JA. Darbepoetin alfa for anemia in patients with low or intermediate-1 risk myelodysplastic syndromes and positive predictive factors of response. Curr Med Res Opin. 2011 May;27(5):951-60. doi: 10.1185/03007995.2011.561834. Epub 2011 Mar 7. PMID 21381892